CLINICAL TRIAL: NCT07146321
Title: A Randomized, Double-blinded, Placebo-controlled Study to Investigate the Effect of a Multivitamin, Multi-nutrient Supplement on Mental and Emotional Wellbeing in Females Aged 43 - 55 Years
Brief Title: A Study to Investigate the Effect of a Multivitamin, Multi-nutrient Supplement on Mental and Emotional Wellbeing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biologica Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AFCRO-196
Record Dates: First submitted 2025-08-08; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Menopause
MeSH Terms: interventions — Geritol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multi-vitamin, multi-nutrient supplement (Active Comparator)
  Interventions: Dietary Supplement: multi-vitamin, multi-nutrient
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: multi-vitamin, multi-nutrient — A multi-vitamin, multi-nutrient combination of approved and/or GRAS ingredients
  Arms: multi-vitamin, multi-nutrient supplement
Dietary Supplement: Placebo — placebo
  Arms: placebo

SUMMARY:
This is a randomized, double-blinded, parallel, placebo-controlled study to investigate the effect of a multivitamin, multi-nutrient supplement on mental and emotional wellbeing in healthy females aged 43 to 55 years, experiencing peri-menopausal and menopausal symptoms

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent.
2. Be between 43 and 55, inclusive.
3. Experiencing a score of >4 on 3 of the symptoms below, within the past 12-months, measured by the MenQoL at Visit 1.

   1. feeling anxious or nervous
   2. difficulty sleeping
   3. feeling tired or worn out
   4. being impatient with other people
4. Ability to wear and interact with a wearable device (ring) for biomarker tracking.
5. Has a minimum 7 days of Oura ring data
6. Willing to consume the Study Product daily for the duration of the study.

Exclusion Criteria:

1. Participants who are pregnant or wish to become pregnant during the study or who are lactating and/or currently breastfeeding.
2. Participants currently of biological childbearing potential, but not using a continuous effective method of contraception, as outlined below:

   1. Complete abstinence from intercourse two weeks prior to administration of the Study Product, throughout the clinical study, until the completion of follow-up procedures or for two weeks following discontinuation of the Study Product in cases where Participant discontinues the study prematurely. (Participants utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding two weeks when they present to the clinic for the final visit).
   2. Has a male sexual partner who is surgically sterilized prior to the Screening Visit and is the only male sexual partner for that Participant.
   3. Sexual partner(s) is/are exclusively female.
   4. Use of acceptable method of contraception, such as a spermicide, mechanical barrier (e.g., male condom, female diaphragm), or tubal ligation. The Participant must be using this method for at least one week prior to and one week following the end of the study.
   5. Use of any non-hormonal intrauterine device (IUD). The Participant must have the device inserted at least two weeks prior to the first screening visit, throughout the study, and two weeks following the end of the study.
3. Drinks more than nationally recommended units of alcohol per day/week. (Defined as <7 standard drinks per week, spread out over the week, with 2 to 3 alcohol-free days per week. Drinks no more than 3 standard drinks on any 1 occasion).
4. Has a history of drug and/or alcohol abuse.
5. Smoker
6. Hypersensitivity that would preclude intake of the Study Products
7. Has any significant acute or chronic coexisting health conditions that would prevent them from fulfilling the study requirements, put the Participant at risk or would confound the interpretation of the study results as judged by the investigator on the basis of medical history and routine laboratory test results. Excluded health conditions include:

   1. Uterine fibroids (current or previous 12 months)
   2. Polycystic ovarian syndrome
   3. Psychiatric disorders (e.g. bipolar, schizophrenia)
8. Current or recent (in the past 12-weeks) use of a medication that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results. Prohibited medications include:

   1. Hypnotic-sedative drugs or sleep aids
   2. Psychotropics (e.g., treatment of anxiety, depression, ADHD etc.)
   3. Steroids (inhaled, intravenous, or oral).
9. Current or recent (in the past 1-week) use of prohibited nutritional or non-nutritional supplements that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results. Prohibited supplements include:

   1. Supplements for the support of menopause symptoms (e.g., red clover, wild yam supplements/creams, ginseng, St John's Wort, DHEA supplements, Phytoestrogen supplements, hormone support supplements)
   2. Supplements that contain study product ingredients
   3. Supplements that support mood and sleep
10. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the study.
11. Participants may not be participating in other clinical studies. If the participant has previously taken part in an experimental study, the Investigator must ensure sufficient time has elapsed before entry to this study to ensure the integrity of the results.

Ages: 43 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-04-05 (Estimated)

PRIMARY OUTCOMES:
Psychosocial symptoms associated with menopause | 12 weeks
  Change in mental and emotional symptoms in menopause in the multivitamin, multi-nutrient supplement group compared to Placebo. Assessed by the Menopause-specific Quality of Life Questionnaire (MenQoL) - psychosocial domain score. Baseline to end of intervention (week 12).

SECONDARY OUTCOMES:
Sexual symptoms of menopause | 12 weeks
  Change in sexual symptoms of menopause (sexual desire, vaginal dryness, and satisfaction) in the multivitamin, multi-nutrient supplement group compared to Placebo. Assessed by the Menopause-specific Quality of Life Questionnaire (MenQoL) - sexual domain score. Baseline to end of intervention (week 12)
Physical symptoms of menopause | 12 weeks
  Change in physical symptoms of menopause (fatigue, sleep disturbances, aches and pains, weight gain, and changes in skin or hair) in the multivitamin, multi-nutrient supplement group compared to Placebo. Assessed by the Menopause-specific Quality of Life Questionnaire (MenQoL) - physical domain score. Baseline to end of intervention (week 12)
Vasomotor symptoms of menopause | 12 weeks
  Change in vasomotor symptoms of menopause (hot flashes, night sweats, and sweating) in the multivitamin, multi-nutrient supplement group compared to Placebo. Assessed by the Menopause-specific Quality of Life Questionnaire (MenQoL) - vasomotor domain score. Baseline to end of intervention (week 12)
Sleep related impairment | 12 weeks
  Change in sleep related impairment (alertness, sleepiness, and tiredness during waking hours) in the multivitamin, multi-nutrient supplement group compared to Placebo. Assessed by the PROMIS® Sleep-Related Impairment - Total Score. Baseline to end of intervention (week 12)
Impact to stress | 12 weeks
  Change in stress in the multivitamin, multi-nutrient supplement group compared to Placebo. Assessed by the DASS-21 - stress score. Baseline to end of intervention (week 12)
Impact to anxiety | 12 weeks
  Change in anxiety in the multivitamin, multi-nutrient supplement group compared to Placebo. Assessed by the DASS-21 - anxiety score. Baseline to end of intervention (week 12)
Impact to working memory | 12 weeks
  Change in memory disturbances in the multivitamin, multi-nutrient supplement group compared to Placebo. Assessed by the Everyday Memory Questionnaire-Revised (EMQ-R) - Total score. Baseline to end of intervention (week 12)
Impact to sleep efficiency | 12 weeks
  Change in sleep quality and patterns in the multivitamin, multi-nutrient supplement group compared to Placebo. Assessed by percentage sleep efficiency, measured using the Oura ring. Baseline to end of intervention (week 12)
Impact to sleep latency | 12 weeks
  Change in sleep quality and patterns in the multivitamin, multi-nutrient supplement group compared to Placebo. Assessed by sleep latency in minutes, measured using the Oura ring. Baseline to end of intervention (week 12)
Impact to total sleep time | 12 weeks
  Change in sleep quality and patterns in the multivitamin, multi-nutrient supplement group compared to Placebo. Assessed by total sleep-in minutes, measured using the Oura ring. Baseline to end of intervention (week 12)
Impact to sleep disturbances | 12 weeks
  Change in sleep quality and patterns in the multivitamin, multi-nutrient supplement group compared to Placebo. Assessed by sleep disturbance as events per hour, measured using the Oura ring. Baseline to end of intervention (week 12)

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Clinical Trials, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No